CLINICAL TRIAL: NCT06586463
Title: Effect Of Kinetic Control Training On Pain And Craniovertebral Angle In Symptomatic Forward Head Posture
Acronym: CairoU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura metwally metwally ali khalifa, asisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005328
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Symptomatic Forwardhead Posture

STUDY DESIGN:
Intervention Model Description: kinetic control training
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Active Comparator): (Control group) receives conventional therapy (cervical, and scapular stabilization exercises, stretching exercises for the pectoralis minor, sternocleidomastoid, scalene muscles and hot pack )
  Interventions: Other: kinitic control training
- kinetic control training (Experimental): takes the same as the control group plus kinetic control. Correction of Low cervical flexion UCM Initially, position the lower and upper cervical spine in neutral with the head supported. the person is trained to perform independent upper cervical flexion (nodding). The upper cervical spine can flex only so far as there is no low cervical flexion. As the ability to control upper cervical extension gets easier and the pattern of dissociation feels less unnatural the exercise can be progressed.
  Correction of scapula and glenohumeral ( UCM) the arm flexion is performed unsupported through the partial range that can be controlled well. This is eventually progressed throughout the full benchmark range with the elbow straight. With visual, auditory and kinaesthetic cues the person becomes familiar with the task of flexing the glenohumeral joint to 90° without scapula movement or glenohumeral translation.
  Interventions: Other: kinitic control training

INTERVENTIONS:
Other: kinitic control training — kinetic control training, Correction of Low cervical flexion UCM Initially, position the lower and upper cervical spine in neutral with the head supported. the person is trained to perform independent upper cervical flexion (nodding). The upper cervical spine can flex only so far as there is no low cervical flexion. As the ability to control upper cervical extension gets easier and the pattern of dissociation feels less unnatural the exercise can be progressed.
  Correction of scapula and glenohumeral ( UCM) the arm flexion is performed unsupported through the partial range that can be controlled well. This is eventually progressed throughout the full benchmark range with the elbow straight. With visual, auditory and kinaesthetic cues the person becomes familiar with the task of flexing the glenohumeral joint to 90° without scapula movement or glenohumeral translation.
  Other Names: conventional treatment

SUMMARY:
The goal of this clinical trial is to investigate the effect of adding kinetic control training of cervical and shoulder joints on pain, neck function, neuromuscular control of the deep cervical flexors, and craniovertebral angle in symptomatic forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) is one of the most common postural deformity, which affects 66% of the patient population with high prevalence among university students due to prolonged usage of computer, smartphones and faulty posture during lectures with lack of awareness about proper posture among them.Participants with FHP exhibited abnormal sensorimotor control and autonomic nervous system dysfunction compared to those with normal head alignment .

Identifying and classifying movement faults is fast becoming the key of recent neuromusculoskeletal rehabilitation. Uncontrolled movement (UCM), contributing to neck pain symptoms, can cause compression or impingement on one side of joints while developing tensile strain on the other side. If UCM is not managed, and the related tissue stress and strain are sustained or repeated beyond the limits of tissue tolerance, multiple tissue pathology may develop eventually and a combination of symptoms may occur . As seen in symptomatic forward head posture.

Along with the identification of site and direction of the faults, direction-movement control intervention(kinetic control) retrains the control of the movement faults. The suggestion is that uncontrolled movement links to the pattern of movement during everyday activities and relates to neck pain. This maneuver can reduce symptoms of neck pain.

ELIGIBILITY:
Inclusion Criteria:

* 1) 50 Subjects of both genders aged 18-40 years old with symptomatic forward head posture (FHP) and Body Mass Index (BMI) less than 30 kg/m2 .

  2) Subjects have FHP if CVA ≤ 50° for assessing FHP 3) Pain between three and eight using numerical pain rating scale NPRS 4) Subjects have non-specific neck pain for at least 3 months

Exclusion Criteria:

* The patients were excluded if they had:

  1. Experienced a history of neck injuries, neck and shoulder surgery
  2. Shoulder trauma, tendinitis, thoracic surgery
  3. Neurological disorders such as cervical spondylosis, spondylolisthesis.
  4. Disc prolapse
  5. Rheumatic disease, fibromyalgia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
craniovertebral angle | up to 4 weeks
  * CVA is defined as the angle formed between a horizontal line through the spinous process of C7 and a line from the tragus of the ear.• To calculate the CVA, reflective markers will be put on the tragus of the ear and the spinous process of C7 before photographing.The eye level will be established by asking the subjects to look forward at a point directly in front of them (colored label will be put on the wall in front of them at their eye level) .
  * A Phone camera will be fixed on an adjustable tripod 1.5 m away from the subject and its base was set at the height of the participant's shoulder. Landmark will be placed on the floor to ensure the same positon of the participants and constant distance from the camera
  * The subjects will be asked to stand comfortably in a normal standing position with their hands hanging beside their bodies and a lateral view picture will be taken from the dominant side by a phone camera. The photos will be analyzed by Kinovea software

SECONDARY OUTCOMES:
neck pain | up to 4weeks
  neck pain by Numerical pain rating scale NPRS . It is a horizontal line with graduation of numbers on it (0-10) 0 means no pain, 10 means the most severe pain that the patient can not tolerate.
neck function | up to 4 weeks
  Neck disability index (Arabic version):
  Assessment of neck function will be performed by Arabic neck disability index. It is a valid and reliable tool in the assessment of neck function . It contains 10 categories. Each category contains six choices (0-5). Score from 0-4 no disability, from 5-15 this is mild, from 15-24 this is moderate, from 25-34 this is severe, more than 34 this is a complete disability
neuromuscular control of the deep cervical flexors (activation and endurance) | up to 4 weeks
  Cranio-cervical flexion test (CCFT): to evaluate neuromuscular control of the deep cervical flexors (activation and endurance) The patient was supine, the head and neck were in a neutral position. The space between the cervical lordotic curve and the table was filled with a pneumatic PBU inflated to 20 mmHg (below the suboccipital region, not below the lower cervical area). The patient performed CCF movement in a graduated approach in 5 increments (22, 24, 26, 28, 30 mmHg), (22, 24, 26, 28, 30 mmHg) that the subject could hold steadily for 10 s using the correct CCF action. Secondly, the assessor evaluated the number of repetitions of a 10 s hold that the patient could perform at their target level. Performance on the CCFT was scored as the pressure level that the patient was able to achieve (activation score) multiplied by the number of repetitions they could perform.

CONTACTS AND LOCATIONS:
Overall Officials: adel rashad ahmed, PhD, Study Chair — professor of physical therapy department of basic science; eman ahmed abdelmoez, PhD, Study Director — professor of physical therapy department of basic science; asmaa hossam eldien, PhD, Study Director — lecturer of physical therapy department of basic science cairo university
Locations (2):
- Egypt (2):
  - cairo university- Egypt, Cairo
  - Cairo University, Cairo

REFERENCES:
- [Result] Khosrokiani Z, Letafatkar A, Sokhanguei Y. Long-term effect of direction-movement control training on female patients with chronic neck pain. J Bodyw Mov Ther. 2018 Jan;22(1):217-224. doi: 10.1016/j.jbmt.2017.06.004. Epub 2017 Jun 13. PMID 29332749
- [Result] Khosrokiani Z, Letafatkar A, Gladin A. Lumbar motor control training as a complementary treatment for chronic neck pain: A randomized controlled trial. Clin Rehabil. 2022 Jan;36(1):99-112. doi: 10.1177/02692155211038099. Epub 2021 Sep 2. PMID 34474578
- [Result] Cagnie B, Struyf F, Cools A, Castelein B, Danneels L, O'leary S. The relevance of scapular dysfunction in neck pain: a brief commentary. J Orthop Sports Phys Ther. 2014 Jun;44(6):435-9. doi: 10.2519/jospt.2014.5038. Epub 2014 May 10. PMID 24816504
- [Result] Ashfaq R, Riaz H. Effect of Pressure biofeedback training on deep cervical flexors endurance in patients with mechanical neck pain: A randomized controlled trial. Pak J Med Sci. 2021 Mar-Apr;37(2):550-555. doi: 10.12669/pjms.37.2.2343. PMID 33679948
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33679948/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24816504/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34474578/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29332749/